CLINICAL TRIAL: NCT06433310
Title: Understanding the Efficacy of Dietary Supplement on Fungal Mycobiota in Healthy Volunteers: A Pilot Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-09026469
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Gut Microbiome; Gut Health; Dietary Supplement; L-Phenylalanine; Phenylpropionic Acid
MeSH Terms: interventions — Phenylalanine; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy (Experimental): Participants will receive one bottle of L-Phenylalanine 500 mg Veg Capsule product on Day 0. All subjects will be asked to start taking the supplement on Day 1 continuing until Day 14. They will be asked to take 2x 500 mg capsules in the morning and 1x 500 mg capsule in the evening daily for 14 days.
  Interventions: Drug: L-Phenylalanine 500 mg Veg Capsule product

INTERVENTIONS:
Drug: L-Phenylalanine 500 mg Veg Capsule product — 500 mg Veg Capsule product

SUMMARY:
The purpose of this study is to explore how the dietary supplement L-Phenylalanine affects the production of the metabolite phenylpropionic acid (PPA) and changes fungal populations of the gut microbiome.

DETAILED DESCRIPTION:
The human gastrointestinal tract hosts a diverse microbial community that has a role in influencing the host's pathophysiological responses. Although there is an abundance of metagenomic data available, the functional dynamics of the gut microbiota still need exploration in different conditions. The microbiota produces various metabolites from dietary products, impacting both host health and pathophysiological functions. The metabolites produced by different microbiota may selectively suppress or stimulate the growth of some components of the gut microbiome, ultimately influencing the dynamic of gut bacterial and fungal populations. Our lab is specifically interested in a metabolite, known as phenylpropionic acid (PPA) produced by a human gut resident bacteria known as Clostridium sporogenes. C. sporogenes produces PPA by metabolizing the amino acid, L-phenylalanine, which is sourced from human diet. Many studies have observed the antimicrobial and antifungal effects of PPA. Our lab determined PPA holds antifungal activity of PPA in the gut of mice colonized with Candida albicans. We are interested in investigating how diversity in the mycobiota populations, which focuses on the fungi species in the human gut, are related to changes in PPA levels.

Therefore, this study will asses whether additional oral supplementation of L-phenylalanine has an effect on the way gut mycobiota responds to this amino acid. Healthy subjects received a 14-day supply of L-phenylalanine supplements and provided stool and blood samples to the study team.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults over the age of 18 years

Exclusion Criteria:

* History of a diagnosis of any gastrointestinal condition, such as inflammatory bowel syndrome or disease
* Antibiotic usage within the past two weeks
* Antifungal usage within the past month
* Allergy to L-Phenylalanine or individuals with phenylketonuria (PKU)
* Adults taking medications known to interact with L-phenylalanine supplements, such as Monoamine Oxidase Inhibitors (MOAI), L-DOPA, and some antipsychotic drugs (complete and extensive drug list will be provided to interested participants during screening)
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in phenylpropionic acid levels from baseline in subject fecal material | Baseline, Week 2 (Day 14)
  Metabolite phenylpropionic acid levels will be measured using mass spectrometry before (baseline) and after intervention
Change in fungal population levels, specifically gut Candida levels, from baseline in subject fecal material | Baseline, Week 2 (Day 14)
  Fungal populations, including Candida, will be measured using microbiota sequencing before (baseline) and after intervention. The most abundant fungal populations will be reported; however, the identity of those populations won't be known until sample analysis.
Change in the number of T cells that react to fungal antigens from baseline in subject blood samples | Baseline, Week 2 (Day 14)
  Blood will be processed through ELISA-based and in vitro restimulation assays to measure T cell reactivity to fungal antigens

SECONDARY OUTCOMES:
Change in phenylpropionic acid levels from baseline in subject fecal material | Baseline, Week 4 (Day 28)
  Metabolite phenylpropionic acid levels will be measured using mass spectrometry before (baseline) and after intervention
Change in fungal population levels, specifically gut Candida levels, from baseline in subject fecal material | Baseline, Week 4 (Day 28)
  Fungal populations, including Candida, will be measured using microbiota sequencing before (baseline) and after intervention. The most abundant fungal populations will be reported; however, the identity of those populations won't be known until sample analysis.
Change in the number of T cells that react to fungal antigens from baseline in subject blood samples | Baseline, Week 4 (Day 28)
  Blood will be processed through ELISA-based and in vitro restimulation assays to measure T cell reactivity to fungal antigens

CONTACTS AND LOCATIONS:
Overall Officials: Iliyan D Iliev, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Belfer Research Building, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No